CLINICAL TRIAL: NCT01766427
Title: Electroacupuncture for Hypertension Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: YueYiDeng (Other)
Responsible Party: Sponsor-Investigator, YueYiDeng, Director of Department of Nephrology of Longhua hospital, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Other Study IDs: 2012LCSY026
Record Dates: First submitted 2013-01-06; First posted 2013-01-11 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: HYPERTENSION RENAL
MeSH Terms: conditions — Hypertension, Renal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- morning electroacupuncture with pills
- afternoon EA with pills
- no EA group with pills

SUMMARY:
1. To observe the Efficiency of Electroacupuncture for Hypertension Patients With Chronic Kidney Disease.
2. To observe if different-time treatment having an impact on Hypertension Patients With Chronic Kidney Disease.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patients with Hypertension

Exclusion Criteria:

* renal replacement therapy
* heart failure
* severe valvular disease
* sustained arrhythmias
* secondary hypertension excluded from renovascular hypertension
* acute cardiovascular events
* infection

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: in the ward of the department of nephrology
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
24 hours Ambulatory Blood Pressure Monitoring Mean arterial pressure change of participants | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Longhua hopsital, Shanghai, Shanghai Municipality, China